CLINICAL TRIAL: NCT06770907
Title: Genetic Carbohydrate Maldigestion As a Model to Study Food Hypersensitivity Mechanism and Guide Personalised Treatment Using a Non-invasive Multiparametric Test (WORK PACKAGE 2)
Brief Title: Genetic Carbohydrate Maldigestion As Model to Study Food Hypersensitivity Mechanism (WORK PACKAGE 2)
Acronym: GenMalCarb2
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: cic bioGune (Unknown); Institute for Clinical Molecular Biology, Christian-Albrechts-University, Kiel (Unknown); University of Veterinary Medicine Hannover (Unknown)
Responsible Party: Principal Investigator, Maura Corsetti, Associate Professor of Gastroenterology, University of Nottingham
Other Study IDs: FMHS 215-0624
Record Dates: First submitted 2024-11-21; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Sucrase Isomaltase Deficiency
Keywords: sucrose isomaltase deficiency
MeSH Terms: conditions — Sucrase-isomaltase deficiency, congenital | interventions — Blood Specimen Collection; Defecation; Magnetic Resonance Imaging; Breath Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, stools and blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Congenital Sucrase-Isomaltase Deficiency: Subjects with congenital sucrase-isomaltase deficiency (CSID) who report symptoms
  Interventions: Other: Blood, stool and saliva collection; Other: Questionnaire completion; Diagnostic Test: Magnetic Resonance Imaging (MRI) and Breath test
- Healthy subjects: Subjects without CSID
  Interventions: Other: Blood, stool and saliva collection; Other: Questionnaire completion; Diagnostic Test: Magnetic Resonance Imaging (MRI) and Breath test
- Asymptomatic controls single carriers: Subjects single carriers for sucrose isomaltase deficiency without symptoms
  Interventions: Other: Blood, stool and saliva collection; Other: Questionnaire completion; Diagnostic Test: Magnetic Resonance Imaging (MRI) and Breath test
- Asymptomatic controls double carriers: Subjects double carriers for sucrose isomaltase deficiency without symptoms
  Interventions: Other: Blood, stool and saliva collection; Other: Questionnaire completion; Diagnostic Test: Magnetic Resonance Imaging (MRI) and Breath test

INTERVENTIONS:
Other: Blood, stool and saliva collection — Blood, stool and saliva collection
Other: Questionnaire completion — Questionnaire on:
  * Hospital Anxiety and Depression Score (HADS) for adults
  * Total glucose and fructose and excess fructose, lactose, sorbitol, mannitol, oligosaccharides (Fructans and GOS) as measured by CNAQ questionnaire for adults and children
  * Patient Health Questionnaire 12 (PHQ-12) Somatic Symptom scale
Diagnostic Test: Magnetic Resonance Imaging (MRI) and Breath test — MRI scans and breath test samples collected after drink test with sucrose

SUMMARY:
Irritable bowel syndrome (IBS) affects one in seven people with gastrointestinal (GI) symptoms that are detected without an established underlying organic cause. IBS strongly impacts quality of life, is a leading cause of work absenteeism, and consumes 0.5% of the healthcare annual budget. It manifests in women more than men with symptoms including abdominal pain, bloating, constipation (IBS-C), diarrhoea (IBS-D), and mixed presentations (IBS-M). The development of therapeutic options is hampered by the heterogeneity of IBS, the lack of specificity of its symptom-based definitions, and the poor understanding of the underlying pathophysiological mechanisms.

Many people with IBS find that certain foods (particularly carbohydrates) trigger their symptoms and avoiding such foods has been shown to be effective in IBS. An example of such a diet is the low-FODMAP (fermentable oligo-, di-, monosaccharides and polyols) exclusion diet, developed by researchers at Monash University. This has suggested that the food-symptom relation may involve malabsorption of carbohydrates due to inefficient enzymatic breakdown of polysaccharides. However, only a percentage of subjects respond to this diet. Overall, the current findings relating to SI, suggest a strong potential for effective personalized therapeutic (dietary) interventions in subgroups of IBS subjects and suggest similar mechanisms should be investigated in relation to other genes involved in the digestion and absorption of carbohydrates (CDGs). This project aims to understand what the mechanisms for GI symptoms in subjects with these genetic alterations are. Aim of the study is to assess the gut response to a sucrose challenge in single-and double-carriers of the common hypomorphic sucrase-isomaltase variant p. (Val15Phe) vs non- carriers (negative controls) and CSID subjects (positive controls), applying an MRI multiparametric test combined with a breath test.

ELIGIBILITY:
Inclusion Criteria for CSID subjects:

* Aged ≥18 (all groups)
* Subjects with genetically proven CSID
* Previous negative endoscopy with biopsies excluding IBD or microscopic colitis in people above 50 years old.
* Negative relevant additional screening (including exclusion of coeliac disease with TTG and IgA)
* Ability to conform to the study protocol including the sucrose challenge.

Exclusion Criteria for CSID subjects:

* Subjects on opioids and use of drugs known to alter GI motility for the duration of the study.
* Presence of concurrent organic gastrointestinal disease (inflammatory bowel disease, coeliac disease, cancer), or a major disease such as diabetes, uncontrolled thyroid disease
* Any history of bowel surgery (not appendectomy or cholecystectomy)
* Contraindication to MRI scanning
* Having taken part in another interventional research study within 3 months
* Concurrent major confounding condition (e.g. alcohol or substance abuse in the last 2 years) based on the study clinician's judgement.

Inclusion Criteria for healthy participants:

* Aged ≥18 years
* Absence of Rome III IBS criteria
* Non-SI variant confirmed (group 1) or Single-SI variants confirmed (group 2) or Double - SI variants confirmed (group 3)
* Ability to conform to the study protocol including the sucrose challenge

Exclusion Criteria for healthy participants:

* Person presenting with a functional or organic GI disorder.
* Person presenting with underlying disease that may involve the GI tract (e.g. Parkinson's disease) or be associated with GI symptoms (e.g. anorexia nervosa, major depression).
* Any history of bowel surgery (not appendectomy or cholecystectomy)
* Contraindication to MRI scanning
* Having taken part in another interventional research study within 3 months
* Concurrent major confounding condition (e.g. alcohol or substance abuse in the last 2 years) based on the clinician's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Single-centre study. CSID subjects will be identified and recruited either with the help of the PPI group through advertisements on social media or flyers at Clinical Genetics and Genomic Conferences and Adult Metabolic Disorder Conferences.
  Healthy participants will be recruited through social media advertisements and posters.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Area under the curve | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
  Area under curve (AUC) of the change from baseline for the MRI measured small bowel water content after the drink test with sucrose

SECONDARY OUTCOMES:
Habitual diet questionnaire | during 4 days before the MRI study
  subject will report food eaten at each meal
MRI measured colon free water content | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
  MRI measured colon free water content, (in arbitrary units) after the drink test
MRI measured small bowel and colon gas content | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
  small bowel and colon gas content (in arbitrary units) after the drink test
MRI measured small bowel and colon volume | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
  small bowel and colon volume in arbritary units after drink test
MRI measured oro-caecal transit time | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
  oro-caecal transit time (OCTT), (in arbitrary units) after the drink test
Breath hydrogen and methane concentration measured in parts per million after drink test | baseline and then 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
Symptoms of nausea, gas/flatulence, bloating and pain/discomfort measured using a Composite Symptom Score after the drink test | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
Total glucose and fructose and excess fructose, lactose, sorbitol, mannitol, oligosaccharides (Fructans and GOS) as measured by Comprehensive Nutrition Assessment Questionnaire | time 0
  CNAQ questionnaires results
Hospital Anxiety and Depression Score | time 0
  scale measuring the score of anxiety and depression
The Patient Health Questionnaire 12 | Time 0
  Scale measuring the psychosomatic score
Stool microbiota taxonomic | Up to 3 days before the MRI study
  Analysis of of microbiota taxonomic in the two stool samples collected by patient during the day before the MRI study day
Stool microbiota alpha and beta diversity measurements | Up to three days before the MRI study day
  Analysis of alfa and beta diversity of microbiota in the two stool samples collected by patient before the study day
Serum levels of short chain fatty acids | At baseline and 0, 60, 120, 180, 240, 300 minutes after the drink test
  Serum levels
Circulating blood glucose levels | Baseline and then 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, 300 minutes after the drink test
Serum levels of surrogates of intestinal permeability (occludin, lipopolysaccharide binding protein) | At baseline and 0, 60, 120, 180, 240, 300 minutes after the drink test
  Serum levels
Serum levels of lipidome and free fatty acids | At baseline and 0, 60, 120, 180, 240, 300 minutes after the drink test
  Serum levels
Serum levels of total serum N-glycome and glucose | At baseline and 0, 60, 120, 180, 240, 300 minutes after the drink test
  Serum levels
Food and drink avoidance questionnaire | at time 0
  patients will respond to the below questions:
  * Name of the food or drink you try to avoid.
  * Please tell us if you try to avoid this food or drink partially or completely? Approximately how long you have tried to avoid this food or drink partially or completely.
  Why do you try to avoid this food or drink partially or completely (including if you have been told to avoid it by a health care professional such as a doctor or dietitian)
Leeds Food Preference Questionnaire | at time 0
  The LFPQ consists of two tasks requiring different interaction from the participant. One task requires an explicit evaluation of each food item using visual analogue scales. The other requires a quick choice to be made between paired combinations of foods. The order of task completion is randomised.
Food Craving Questionnaire - State (FCQ-S) | at time 0
  participants respond to 14 questions about sugary food and they will respond with a scale from 1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Corsetti, Medical Doctor, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No